CLINICAL TRIAL: NCT04001647
Title: Targeting Endoplasmic Reticulum Stress in Aging- and Obesity-Induced Vascular Dysfunction
Brief Title: Targeting ER Stress in Vascular Dysfunction
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: IRB approval has been withdrawn
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TUDCA and Vascular Health
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-07

CONDITIONS: Vasodilation; Arterial Stiffness
Keywords: ER stress; Unfolded protein response; Vascular function; Aging; Obesity; TUDCA
MeSH Terms: conditions — Aneurysm; Obesity | interventions — Acetylcholine; Nitroprusside; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Participants from each group (young healthy weight, young obese, older healthy weight, older obese) will be studied before and after 8 weeks of tauroursodeoxycholic acid (TUDCA) treatment. Additional older obese participants will be studied before and after 8 weeks of a placebo treatment.
Who Masked: Participant, Investigator
Masking Description: A study monitor not involved in data collection or analysis will perform masking of both the participant and investigator for the interventions for the older obese participants. These participants will be randomized into placebo or TUDCA treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TUDCA (Experimental): Young and older healthy weight and obese participants will visit the lab for assessment of vascular function prior to the intervention. Aortic stiffness will be evaluated non-invasively using carotid-femoral pulse-wave velocity. A physician will place a catheter in the brachial artery for endothelial cell biopsies and local vasodilator infusions. A venous catheter will also be placed for the systemic ascorbic acid infusion. Aortic stiffness measures and vascular responses to vasodilator infusions will be performed before and after the ascorbic acid infusion. Following the completion of the vascular assessments, participants will receive 1750 mg/day of the dietary supplement tauroursodeoxycholic acid (TUDCA) for 8 weeks. Participants will return to the lab after the 8 week intervention and the vascular assessments described above will be repeated.
  Interventions: Drug: Acetylcholine; Drug: Sodium Nitroprusside; Drug: Ascorbic Acid
- Placebo (Placebo Comparator): Older obese participants will visit the lab for assessment of vascular function prior to the intervention. Aortic stiffness will be evaluated non-invasively using carotid-femoral pulse-wave velocity. A physician will place a catheter in the brachial artery for endothelial cell biopsies and local vasodilator infusions. A venous catheter will also be placed for the systemic ascorbic acid infusion. Aortic stiffness measures and vascular responses to vasodilator infusions will be performed before and after the ascorbic acid infusion. Following the completion of the vascular assessments, participants will receive oral capsules containing a placebo treatment for 8 weeks. Participants will return to the lab after the 8 week intervention and the vascular assessments described above will be repeated.
  Interventions: Drug: Acetylcholine; Drug: Sodium Nitroprusside; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Acetylcholine — Endothelium-dependent vasodilation will be determined via graded intra-arterial infusions of acetylcholine (ACh). Doses of 1, 4, 8, and 16 μg/100ml forearm volume/min will be infused in the brachial artery for 3 minutes each.
  Other Names: ACh
Drug: Sodium Nitroprusside — Endothelium-independent vasodilation will be determined via graded intra-arterial infusions of sodium nitroprusside (SNP). Doses of 0.25, 0.5, 1, and 2 μg/100ml forearm volume/min will be infused in the brachial artery for 3 minutes each.
  Other Names: SNP
Drug: Ascorbic Acid — The influence of oxidative stress on arterial stiffness and vasodilation will be assessed by using intravenous ascorbic acid (AA). A single supra-physiological dose of 0.06 g/kg fat-free mass (FFM) will be infused over 20 min followed by a drip infusion of 0.02 g/kg FFM administered over 60 min.
  Other Names: AA; Vitamin C

SUMMARY:
Aging and obesity are both risk factors for cardiovascular disease (CVD). One process that links both of these conditions to CVD is vascular dysfunction. Data from animal studies indicate that endoplasmic reticulum (ER) stress may play an important role in the development of endothelial dysfunction in aging and obesity. Therefore, the goal of this study is to investigate the relative contributions of aging and obesity on vascular dysfunction and ER stress. Additionally, this study will determine if taking an oral supplement for 8 weeks will improve vascular dysfunction and ER stress. Results from this study have the potential to identify a safe treatment option for improving vascular function in aging and obese populations.

DETAILED DESCRIPTION:
Aging is the primary risk factor for cardiovascular disease (CVD). One critical process that links aging to CVD is the development of vascular dysfunction, characterized by endothelial dysfunction and arterial stiffness. Both endothelial dysfunction and arterial stiffness predict cardiovascular events in older individuals. Aging often coincides with obesity, another independent risk factor for CVD. Although vascular function is well characterized in both aging and obesity, it's unclear how these two conditions interact to modulate vascular function, and whether the combination of aging and obesity has additive or compounding effects on endothelial dysfunction and arterial stiffness.

Currently, it is unknown whether vascular dysfunction is driven by the same underlying cellular mechanisms in aging and obesity. Accumulating data in experimental animals suggest that ER stress may be an important factor in aging- and obesity-related vascular dysfunction. Additionally, middle-aged and older obese adults with endothelial dysfunction display evidence of ER stress within biopsied endothelial cells. In light of these data, the overall goal of this proposal is to test the hypothesis that ER stress is associated with human vascular dysfunction in the settings of aging and obesity, and to determine the efficacy of the chemical chaperone tauroursodeoxycholic acid (TUDCA), an established inhibitor of ER stress, to reduce endothelial cell ER stress and improve vascular function in these at-risk individuals. Results from this study have the potential to identify a novel, safe, and clinically relevant intervention strategy for the treatment of vascular dysfunction in an aging population at high-risk for the development of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy weight adults (age: 18-35; BMI 18.5-24.9 kg/m2)
* Young, obese adults (age: 18-35; BMI 30- 39.9 kg/m2)
* Older, healthy weight adults (age: 60-80; 18.5-24.9 kg/m2)
* Older, obese adults (age: 60-80; 30-39.9 kg/m2)

Exclusion Criteria:

* blood pressure >140/90 mmHg
* triglycerides >500 mg/dL or LDL cholesterol >190 mg/dL
* current smoking or history of smoking in the last 12 months
* diagnosed chronic disease including cancer, cardiovascular, diabetes, kidney, liver, and pancreatic disease
* weight change >3 kg in the past 3 months or actively trying to lose weight
* >12 alcoholic drinks/week
* hormone replacement therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent vasodilation | Change in baseline vasodilation at 8 weeks
  Blood flow response to increasing doses of acetycholine
Endothelium-independent vasodilation | Change in baseline vasodilation at 8 weeks
  Blood flow response to increasing doses of sodium nitroprusside
Aortic stiffness | Change in baseline pulse-wave velocity at 8 weeks
  Carotid-femoral pulse-wave velocity
Endothelial cell ER stress marker ATF6 | Change in baseline endothelial ATF6 at 8 weeks
  Protein expression of activating transcription factor 6 (ATF6)
Endothelial cell ER stress marker PERK | Change in baseline endothelial PERK at 8 weeks
  Protein expression of RNA-dependent protein kinase- like ER eukaryotic initiation factor-2α kinase (PERK)
Endothelial cell ER stress marker IRE1α | Change in baseline endothelial IRE1α at 8 weeks
  Protein expression of inositol-requiring ER-to-nucleus signaling protein 1(IRE1α)
Endothelial cell ER stress marker CHOP | Change in baseline endothelial CHOP at 8 weeks
  Protein expression of CCAAT-enhancer-binding protein homologous protein (CHOP)
Endothelial cell ER stress marker GRP78 | Change in baseline endothelial GRP78 at 8 weeks
  Protein expression of glucose-regulated protein 78 (GRP78)
Endothelial cell ER stress marker GADD34 | Change in baseline endothelial GADD34 at 8 weeks
  Protein expression of growth arrest and DNA damage-inducible 34 (GADD34)
Endothelial cell oxidative stress marker p47phox | Change in baseline endothelial p47phox at 8 weeks
  Protein expression of nicotinamide adenine dinucleotide phosphate (NADPH) oxidase subunit p47phox
Endothelial cell oxidative stress marker NT | Change in baseline endothelial NT at 8 weeks
  Protein expression of nitrotyrosine (NT)
Endothelial cell oxidative stress marker MnSOD | Change in baseline endothelial MnSOD at 8 weeks
  Protein expression of manganese superoxide dismutase (MnSOD)
Endothelial cell oxidative stress marker CuZnSOD | Change in baseline endothelial CuZnSOD at 8 weeks
  Protein expression of copper-zinc SOD (CuZnSOD)
Endothelial cell inflammatory marker p65 | Change in baseline endothelial p65 at 8 weeks
  Protein expression of nuclear factor kappa B phosphorylated p65 subunit
Endothelial cell inflammatory marker IκBα | Change in baseline endothelial IκBα at 8 weeks
  Protein expression of phosphorylated inhibitor of kappa B (IκBα)
Endothelial cell inflammatory marker TNFα | Change in baseline endothelial TNFα at 8 weeks
  Protein expression of tumor necrosis factor-alpha (TNFα)
Endothelial cell inflammatory marker IL-6 | Change in baseline endothelial IL-6 at 8 weeks
  Protein expression of interleukin-6 (IL-6)

SECONDARY OUTCOMES:
Circulating glucose | Change in baseline blood glucose at 8 weeks
  Blood glucose
Circulating insulin | Change in baseline insulin at 8 weeks
  Blood levels of insulin
Circulating cholesterol | Change in baseline total cholesterol, LDL cholesterol, and HDL cholesterol at 8 weeks
  Blood levels of total cholesterol, LDL cholesterol, and HDL cholesterol
Circulating triglycerides | Change in baseline triglycerides at 8 weeks
  Blood levels of triglycerides
Circulating CRP | Change in baseline CRP at 8 weeks
  Blood levels of C-reactive protein (CRP)
Circulating IL-6 | Change in baseline IL-6 at 8 weeks
  Blood levels of interleukin (IL)-6
Circulating IL-18 | Change in baseline IL-18 at 8 weeks
  Blood levels of interleukin (IL)-18
Circulating IL-10 | Change in baseline IL-10 at 8 weeks
  Blood levels of interleukin (IL)-10
Circulating IL-1β | Change in baseline IL-1β at 8 weeks
  Blood levels of interleukin (IL)-1 beta (β)
Circulating TNFα | Change in baseline TNFα at 8 weeks
  Blood levels of tumor necrosis factor-alpha (TNFα)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Dinenno, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No